CLINICAL TRIAL: NCT06328400
Title: A Multiple-dose, Randomized, Double-blind, Placebo-controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral Deuremidevir Hydrobromide for Suspension in Chinese Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral Deuremidevir Hydrobromide for Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VV116-RSV-02
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Suspensions; GS-621763

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Deuremidevir Hydrobromide for Suspension 900mg group, twice a day (Experimental): 9 subjects will receive Deuremidevir Hydrobromide for Suspension 900mg, orally, Q12h, 5.5 days; 3 subjects will receive Deuremidevir Hydrobromide for Suspension Placebo 900mg, orally, Q12h, 5.5 days.
  Interventions: Drug: Deuremidevir Hydrobromide for Suspension; Drug: Deuremidevir Hydrobromide for Suspension Placebo
- Deuremidevir Hydrobromide for Suspension 900mg group, 3 times a day (Experimental): 9 subjects will receive Deuremidevir Hydrobromide for Suspension 900mg, orally, Q8h, 5.5 days; 3 subjects will receive Deuremidevir Hydrobromide for Suspension Placebo 900mg, orally, Q8h, 5.5 days.
  Interventions: Drug: Deuremidevir Hydrobromide for Suspension; Drug: Deuremidevir Hydrobromide for Suspension Placebo
- Deuremidevir Hydrobromide for Suspension 1200mg group, twice a day (Experimental): 9 subjects will receive Deuremidevir Hydrobromide for Suspension 1200mg, orally, Q12h, 5.5 days; 3 subjects will receive Deuremidevir Hydrobromide for Suspension Placebo 1200mg, orally, Q12h, 5.5 days.
  Interventions: Drug: Deuremidevir Hydrobromide for Suspension; Drug: Deuremidevir Hydrobromide for Suspension Placebo

INTERVENTIONS:
Drug: Deuremidevir Hydrobromide for Suspension — Experimental: Deuremidevir Hydrobromide for Suspension 900mg group, twice a day Experimental: Deuremidevir Hydrobromide for Suspension 900mg group, 3 times a day Experimental: Deuremidevir Hydrobromide for Suspension 1200mg group, twice a day
  Other Names: VV116
Drug: Deuremidevir Hydrobromide for Suspension Placebo — Experimental: Deuremidevir Hydrobromide for Suspension 900mg group, twice a day Experimental: Deuremidevir Hydrobromide for Suspension 900mg group, 3 times a day Experimental: Deuremidevir Hydrobromide for Suspension 1200mg group, twice a day
  Other Names: VV116 Placebo

SUMMARY:
This trial is a multi dose, randomized, double-blind, placebo-controlled, single center Phase I clinical study. The purpose of this study is to evaluate the safety, tolerability, and PK characteristics of Deuteromide Hydrobromide for Suspension administered multiple times in healthy volunteers.

DETAILED DESCRIPTION:
Two groups are initially set up, starting from Group 1 and progressing sequentially to Group 2. After all volunteers in the first group (900 mg BID group) complete the safety follow-up on the 4th day after the last dose (i.e. D10), the safety information and PK data will be reviewed jointly by the researchers and sponsors before the second group of volunteers starting administration. The preferred dose for the second group is 900 mg TID, and if there are safety risks found after the Group 1 study, it will be adjusted to 1200 mg BID or other appropriate dosage and frequency.

A total of 24 volunteers are planned to be enrolled, with 12 volunteers in each group. The trial drug and placebo will be allocated in a 3:1 ratio, with 9 volunteers in each group receiving the trial drug and 3 volunteers receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 45 years old, males or females;
2. Body weight no less than 45 kg, Body Mass Index of 18 to 25 kg/m2;
3. Vital signs examination, physical examination, laboratory examination and electrocardiogram examination results were normal or abnormal without clinical significance;
4. Subjects who are willing to take proper contraceptive during the study and within 3 months after the last administration;
5. Subjects who are able to understand and follow the study plans and instructions; Subjects who have voluntarily decided to participate in this study, and signed the informed consent form.

Exclusion Criteria:

1. Subjects with hypersensitivity to deuremidevir hydrobromide for suspension or any of the excipients;
2. Subjects with allergic diseases or allergic constitution;
3. Subjects with central nervous system, cardiovascular system,gastrointestinal, respiratory system, urinary, Hematologic System,metabolic disorders that require medical intervention or other diseases(such as psychiatric history) that are not suitable for clinical trials;
4. Subjects with acute upper respiratory tract infection within 2 weeks before screening;
5. Subjects who have received blood transfusion or used blood products within 3 months before screening or who have lost more than ≥400 mL of blood due to other reasons (except female physiological blood loss);
6. Subjects who have participated in clinical trials of other drugs within 90 days before screening;
7. Subjects who have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health products within 2 weeks before screening;
8. Subjects who have consumed grapefruits, pomelos, oranges, etc. within the previous 7 days before screening and do not agree to stop consuming the above fruits and beverages during the trial period;
9. Being a drug addict or alcohol addict within one year before screening,being an alcoholic at present or in the past (drinking more than 14 standard units per week, and one standard unit contains 14 g of alcohol,such as 360 mL of beer or 45 mL of strong liquor with 40% alcohol content or 150 mL of wine), or being positive in the alcohol breath tests;
10. Subjects who smoked more than 5 cigarettes a day within one year before screening;
11. Subjects who can't quit smoking or drinking during the trial period;
12. Subjects who are positive for hepatitis B virus surface antigen, hepatitis C virus antibody, Treponema pallidum antibody (TPPA) or human immunodeficiency virus antibody (Anti-HIV);
13. Abnormal chest X-ray or CT results with clinical significance;
14. Pulse rate>100 beats per minute, or systolic blood pressure ≥ 140 mmHg or<90 mmHg, or diastolic blood pressure ≥ 90 mmHg or<50 mmHg at screening or baseline;
15. Total bilirubin (TBIL) > upper limit of normal value (ULN), Alanine transaminase (ALT) or aspartate transaminase (AST) > 1.5 times ULN at screening or baseline;
16. The glomerular filtration rate (eGFR) < 90 ml/min at screening or baseline;
17. Any of the following blood routine examination results during screening or baseline were lower than the lower limit of normal: white blood cell count, absolute value of lymphocytes, percentage of lymphocytes, percentage of neutrophils, absolute value of neutrophils;
18. Abnormal ECG at screening or baseline, including QTcF (after heart rate correction) >450 ms for males and > 470 ms for females in single examinations, and/or other abnormalities with clinical significance;
19. Pregnant or lactating females, or male volunteers whose spouses have planned pregnancy within 3 months;
20. The investigator believes that there are other unsuitable factors for this volunteer to participate this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From Day1 to Day10 after administration
  Incidence of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
Cmax | 168 hours after administration
  maximum observed plasma concentration
Tmax | 168 hours after administration
  time at which Cmax occurs
AUC0- t | 168 hours after administration
  area under the plasma concentration time curve from time zero to the last quantifiable concentration
AUC0-∞ | 168 hours after administration
  area under the plasma concentration time curve from time zero to infinity
t1/2 | 168 hours after administration
  terminal half life

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojie Wu, Principal Investigator — Hushan Hospital Fudan university
Locations (1):
- Hushan Hospital Fudan university, Shanghai, Shanghai Municipality, China